CLINICAL TRIAL: NCT04974905
Title: Retrograde Approach for Management of Infrainguinal Arterial Occlusive Disease After Failed Antegrade Approach in Critical Limb Ischemia Patients; Feasibility, Safety, and Procedure Related Outcomes.
Brief Title: Retrograde Recanalization of Infrainguinal Arterial Occlusive Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Abdelmagied Ragb Fouda, assistant lecturer in the department of vascular surgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-07-22
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with infrainguinal arterial occlusive disease after failed antegrade approach (Other)
  Interventions: Procedure: retrograde access for re-canalization of infra-inguinal arterial occlusive disease

INTERVENTIONS:
Procedure: retrograde access for re-canalization of infra-inguinal arterial occlusive disease — after failed antegrade approach for re-canalization of infra-inguinal arterial occlusive disease( failed reentry into the distal true lumen), the retrograde approach will be attempted

SUMMARY:
The spectrum of lower extremity peripheral arterial disease (PAD) ranges from exhibiting no symptoms to limb threatening gangrene. The number of patients living with it is rising steadily owing to increased life expectancy, obesity, diabetes, and tobacco consumption.

Critical limb ischemia (CLI) is the terminal and the most serious stage of PAD in which blood flow to the lower extremity does not meet metabolic demands of the tissues at rest. The diagnosis is mainly clinical and patients are presented with rest pain, minimal tissue loss or frank gangrene.

Revascularization strategies include endovascular procedures and surgical bypass.Endovascular therapy has evolved as an attractive, minimally invasive method of revascularization especially in the more frequently encountered patients with medical and anatomical contraindications to surgical revascularization.

Antegrade approach is the standard approach in infrainguinal arterial occlusive disease,however, failure occurs in about 20% of infrainguinal attempts.Retrograde approach is used as a backup technique in failed cases.

ELIGIBILITY:
Inclusion Criteria:

patients with;

1. CLI consistent with Rutherford categories (4-5).
2. Infrainguinal arterial occlusive disease with a patent distal part of at least one tibial vessel runoff to the foot.

Exclusion Criteria:

patients with the following conditions will be excluded:

1. Non-salvageable limbs.
2. Life threatening infections requiring major amputation.
3. Ulcers at the area of intended puncture.

Ages: 35 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
safety of retrograde approach as regard occurrence of procedure specific complications | within one year of follow up
  safety of retrograde approach after failed antegrade approach for recanalization of infrainguinal arterial occlusive disease, in the light of complications which are classified into major or minor according to the reporting standards of society of vascular surgery.this complications will be looked for and data will be collected
feasibility of retrograde approach as regard successful retrograde puncture and technical success after failed antegrade approach for recanalization of infrainguinal arterial occlusive disease. | within one year of follow up
  it means that this approach can be used successfuly in clinical practice and this will be assessd by measuring successful retrograde puncture and technical success.
  successful retrograde puncture means successful performance of retrograde puncture at any of the retrograde distal puncture sites with intraluminal placement of the retrograde guidewire confirmed by contrast angiography without causing procedure specific complications namely local dissection, rupture, or an arteriovenous fistula at puncture site.
  technical success is defined as successful puncture followed by successful crossing of the occlusion and regain of inline flow to the foot with less than 30%residual stenosis after treatment.

SECONDARY OUTCOMES:
clinical success of the procedure | within one year of follow up
  immediate clinical success is defined as regain of distal pulses, revascularization warmness and edema, and/or disappearance of rest pain.
One year limb salvage rate of the procedure | within one year of follow up
  limb salvage is defined as healing of existing wounds with no amputation proximal to metatarsus.

REFERENCES:
- [Background] Mustapha JA, Saab F, McGoff TN, Adams G, Mullins JR, Al-Dadah A, Jaff MR, Goodney PP, Khawaja F, Diaz-Sandoval LJ. Tibiopedal arterial minimally invasive retrograde revascularization (TAMI) in patients with peripheral arterial disease and critical limb ischemia. On behalf of the Peripheral Registry of Endovascular Clinical Outcomes (PRIME). Catheter Cardiovasc Interv. 2020 Feb 15;95(3):447-454. doi: 10.1002/ccd.28639. Epub 2019 Dec 13. PMID 31834669
- [Background] Hendricks NJ, Sabri SS. Subintimal arterial flossing with antegrade-retrograde intervention (SAFARI) and rertograde access for critical limb ischemia. Tech Vasc Interv Radiol. 2014 Sep;17(3):203-10. doi: 10.1053/j.tvir.2014.08.009. Epub 2014 Sep 4. PMID 25241321
- [Background] Bazan HA, Le L, Donovan M, Sidhom T, Smith TA, Sternbergh WC 3rd. Retrograde pedal access for patients with critical limb ischemia. J Vasc Surg. 2014 Aug;60(2):375-81. doi: 10.1016/j.jvs.2014.02.038. Epub 2014 Mar 18. PMID 24650744